CLINICAL TRIAL: NCT05510167
Title: Impact of Post-ablation Alcohol Intake on Arrhythmia Recurrence, Quality of Life and Cognition in Patients With Atrial Fibrillation
Brief Title: Post-ablation Alcohol Impacts Arrhythmia Recurrence, Quality of Life and Cognition in AF
Acronym: PLATINUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TCAI
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: Alcohol; AF; catheter ablation; recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Intervention Model Description: Paroxysmal and Persistent AF patients undergoing their first catheter ablation will be screened for eligibility and those that meet the criteria and consent to participate will be randomly assigned to group 1 or 2.
  Study period will start from the day after the procedure and continue for 8 months (2-month blanking period+ 6 months follow-up).
  Group 1: Complete abstinence or ≤2 drinks/week in group 1 during the study period Group 2: Allowed to continue their pre-ablation drinking habit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Active Comparator): Complete abstinence or ≤2 drinks/week in group 1 during the study period
  Interventions: Behavioral: Study arm
- Control (Active Comparator): Allowed to continue their pre-ablation drinking habit
  Interventions: Behavioral: Study arm

INTERVENTIONS:
Behavioral: Study arm — Participants will be asked to completely abstain from drinking or consume 2 or less drinks per week for 8 months following catheter ablation

SUMMARY:
Earlier studies have shown a dose-dependent relationship between alcohol intake and incident atrial fibrillation (AF) as well as a causal link with several risk factors for AF such as hypertension, obesity and sleep apnea. However, the effect of drinking (alcohol) on post-ablation outcome such as arrhythmia recurrence, quality of life (QoL) and cognitive function in AF patients is unclear. Therefore, we aim to find the answer for a very frequently asked question, "is it safe to continue drinking alcohol (at the pre-ablation level) following catheter ablation OR should the intake be reduced for better outcome?", in this randomized trial.

DETAILED DESCRIPTION:
1. BACKGROUND Earlier studies have not only reported alcohol-abstinence to be associated with lower recurrence of AF in patients receiving non-ablative antiarrhythmic therapy, but also unfavorable outcome among regular drinkers (high frequency and quantity) compared to non-drinkers undergoing AF ablation (1-3). In a meta-analysis of 14 studies, where the effect measures for AF associated with highest vs lowest alcohol intake were pooled for analysis, not consuming alcohol was observed to be the most favorable in terms of AF risk reduction (4). Larsson et al reported alcohol drinking, even in moderate quantity, to be a risk factor for incident AF, whereas Zhang et al observed moderate drinking to be associated with high AF risk in men only and not in females (5, 6). Moreover, a causal link between alcohol intake and other cardiovascular morbidities such as obesity, hypertension, left ventricular dysfunction and sleep apnea that are known risk factors for AF has been documented by several studies (1). Thus, we know that alcohol consumption, even in moderate quantity, increases the risk for AF, although may not be across genders. Observational studies also have shown unfavorable procedure outcome to be more common in drinkers compared to non-drinkers receiving AF ablation. However, there is no randomized data to support the latter statement. Additionally, there are no data on the influence of alcohol intake on the cognitive function and QoL in AF patients receiving catheter ablation. Therefore, this investigator-initiated, randomized trial has been designed to examine the impact of alcohol intake vs abstinence on arrhythmia recurrence and burden, QoL and cognitive function in regular drinkers undergoing their first catheter ablation.
2. STUDY RATIONALE We hypothesize that alcohol-abstinence will significantly improve the procedural outcome, QoL and cognitive function in the study population compared to the non-abstinence cohort.
3. STUDY OBJECTIVES Primary Objective Arrhythmia recurrence across all AF types at 8 months after the ablation procedure, off- or on-antiarrhythmic drug (AAD) Secondary Objective 1) Change in QoL score measured by AFEQT survey at baseline and 6 months 2) Change in cognitive function measured by MoCA survey 3) Arrhythmia burden at follow-up

Study period will start from the day after the procedure and continue for 8 months (2-month blanking period+ 6 months follow-up).

Group 1: Complete abstinence or ≤2 drinks/week in group 1 during the study period Group 2: Allowed to continue their pre-ablation drinking habit

ELIGIBILITY:
Inclusion Criteria:

* AF patients that regularly consume >5 alcoholic drink (*12 g of pure alcohol/drink)/week
* Paroxysmal or persistent AF
* First catheter ablation History of alcohol-induced arrhythmia
* Willing to sign the written informed consent

Exclusion Criteria:

* Binge drinkers (alcohol dependence)
* Non-drinkers
* LVEF <35%
* Psychiatric conditions
* MoCA score ≤ 17 on Montreal Cognitive Assessment (MoCA)
* Patients with established dementia
* Medically unstable patients (acute/unstable or poorly controlled problems that would demand focused, relatively urgent or emergent medical attention)
* Unwilling for alcohol-abstinence
* Long-standing persistence AF
* Patient under legal protection
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia recurrence | 8 months after the ablation procedure for AF
  Arrhythmia recurrence across all AF types at 8 months after the ablation procedure, off- or on-antiarrhythmic drug (AAD)

SECONDARY OUTCOMES:
Change in QoL | 6 months after the blanking period of 2 months
  Change in QoL measured by AFEQT survey at baseline and 6 months
Change in cognitive function | 6 months after the blanking period of 2 months
  Change in cognitive function measured by MoCA survey
Arrhythmia burden | 6-8 months following ablation
  Arrhythmia burden at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, Principal Investigator — Texas Cardiac Arrhythmia Institute, St.

IPD SHARING:
Plan to Share IPD: No